CLINICAL TRIAL: NCT07401394
Title: BAR-TAX - Tranexamic Acid in Bariatric Surgery. Use of Tranexamic Acid and Bleeding Management in Bariatric Surgery: A Prospective Study in a High-Volume Center.
Brief Title: BAR-TAX - Tranexamic Acid in Bariatric Surgery.
Acronym: BAR-TAX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Maria Hospital - GVM Care & Research (Other)
Responsible Party: Principal Investigator, Libero Luca, MD, Santa Maria Hospital - GVM Care & Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GVM_BAR-TAX; BAR-TAX_GVM (Other: Scientific Board GVM)
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bariatric Surgery; Bariatric Patients; Bariatric Surgery Complications; Bleeding; Tranexamic Acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Patients treated with perioperative tranexamic acid will be compared with a historical cohort managed under the previous institutional protocol without TXA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BAR_TAX (Experimental): The TAX arm includes patients undergoing bariatric surgery who receive perioperative tranexamic acid according to the BAR-TAX protocol. Outcomes will be compared with a historical control arm consisting of patients treated under the previous institutional protocol without tranexamic acid administration.
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Tranexamic acid is administered intravenously according to a standardized perioperative regimen. Patients receive 2 g of tranexamic acid diluted in 250 mL of normal saline during anesthetic induction, followed by 2 g intravenously at 8 hours and 12 hours postoperatively. All patients are managed according to standardized perioperative care pathways, including venous thromboembolism prophylaxis and ERABS protocols.

SUMMARY:
Perioperative bleeding is a relevant complication in bariatric surgery and may lead to hemoglobin decrease, blood transfusions, reinterventions, prolonged hospital stay, and increased healthcare costs. Tranexamic acid (TXA), an antifibrinolytic agent, has demonstrated efficacy in reducing surgical bleeding in several surgical specialties, with a favorable safety profile when appropriately used. However, evidence in bariatric surgery remains limited, particularly considering the intrinsically increased thromboembolic risk of obese patients.

The BAR-TAX study is a prospective, single-center study conducted in a high-volume bariatric surgery center, aiming to evaluate the efficacy and safety of perioperative TXA administration compared with standard care without TXA. The primary objective is to assess whether TXA reduces the incidence of clinically significant bleeding within 48-72 hours after bariatric surgery. Secondary objectives include evaluation of hemoglobin drop, transfusion rates, need for hemostatic procedures or reoperation, thromboembolic events, postoperative complications, length of hospital stay, readmissions, and TXA-related adverse events.

DETAILED DESCRIPTION:
Bariatric surgery, including procedures such as Sleeve Gastrectomy, Roux-en-Y Gastric Bypass, Transit Bipartition, and revisional surgery, is associated with a non-negligible risk of perioperative and postoperative bleeding. Clinically significant bleeding may result in adverse outcomes such as increased transfusion requirements, reintervention, prolonged hospitalization, and higher healthcare resource utilization. At the same time, obese patients represent a population at increased baseline risk for venous thromboembolism, requiring careful balancing between bleeding prevention and thromboembolic safety.

Tranexamic acid (TXA) is an antifibrinolytic agent that inhibits plasminogen activation and fibrin degradation, thereby stabilizing clot formation. Its perioperative use has been widely adopted in orthopedic, cardiac, and trauma surgery, with consistent evidence supporting reductions in blood loss and transfusion requirements without a significant increase in thromboembolic events when used according to established protocols. Emerging data in bariatric surgery suggest similar benefits; however, robust prospective data in this specific population are still limited.

The BAR-TAX study is designed as a prospective, non-funded, single-center observational study conducted in a high-volume bariatric surgery unit. Adult patients (≥18 years) with a BMI ≥30 kg/m² undergoing primary or revisional bariatric surgery will be eligible for inclusion. Patients with recent venous thromboembolism, major uncontrolled thrombophilia, severe renal insufficiency, uncontrolled seizure disorders, known TXA allergy, or pregnancy will be excluded.

Patients in the TXA group will receive a standardized perioperative TXA regimen consisting of 2 g administered intravenously during anesthetic induction, followed by 2 g at 8 hours and 2 g at 12 hours postoperatively. All patients will be managed according to standardized perioperative care pathways, including optimized intraoperative hemostasis, venous thromboembolism prophylaxis based on institutional protocols, ERABS principles, and standardized postoperative monitoring.

The primary endpoint is the incidence of clinically significant bleeding within 48-72 hours after surgery, defined by the presence of at least one of the following: hemoglobin drop ≥2 g/dL associated with clinical signs, need for blood transfusion, bleeding requiring endoscopic, radiologic, or surgical intervention, or hemodynamic instability attributable to bleeding. Secondary endpoints include hemoglobin variation at 24 and 72 hours, estimated hidden blood loss, transfusion rate and indications, need for reintervention or hemostatic procedures, 30-day venous thromboembolic events, postoperative complications classified according to Clavien-Dindo, length of hospital stay, readmissions, and TXA-related adverse events such as seizures or allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Both sexes
* BMI ≥30 kg/m²
* Candidates for primary or revisional bariatric surgery

Exclusion Criteria:

* Recent history of DVT/PE (e.g., <12 months) or major thrombophilia not adequately managed
* Severe renal insufficiency (e.g., eGFR <30 mL/min/1.73 m²) or need for unmanageable dose adjustment
* History of uncontrolled seizures/epilepsy (dose-dependent risk)
* Known allergy to TXA
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
TAX and bleeding in bariatric surgery | 12 months
  To evaluate whether perioperative TAX use reduces the incidence of clinically significant bleeding within 48-72 hours after surgery (defined as at least one of the following: hemoglobin drop ≥2 g/dL with clinical signs, need for transfusion, bleeding requiring a procedure/endoscopy/surgery, hemodynamic instability attributable to bleeding).

SECONDARY OUTCOMES:
Hidden blood loss | 12 months
  Reduction in hemoglobin drop at 24 h and 72 h (ΔHb) and estimation of hidden blood loss.
Transfusion rate | 12 months
  Transfusion rate (units of packed red blood cells) and indication.
Rate of re-operation | 12 months
  Rate of re-operation/hemostatic revision or hemostatic procedures (endoscopy/interventional radiology).
Incidence of complications | 12 months
  Incidence of venous thromboembolic events at 30 days. Incidence of complications at 30 days (Clavien-Dindo classification, late hemorrhagic complications).
Hospital stay | 12 months
  Length of hospital stay and readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Braun, MD, Principal Investigator — GVM Care & Research
Locations (1):
- Santa Maria Hospital - GVM, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 't Hart JWH, Noordman BJ, Wijnand JMA, Biter LU, Verbrugge SJC, Birnie E, Dunkelgrun M, Huisbrink J, Apers JA. Peroperative administration of tranexamic acid in sleeve gastrectomy to reduce hemorrhage: a double-blind randomized controlled trial. Surg Endosc. 2023 Oct;37(10):7455-7463. doi: 10.1007/s00464-023-10232-5. Epub 2023 Jul 3. PMID 37400687
- [Background] Bieniaszewski K, Proczko-Stepaniak M, Wilczynski M, Nowicki P, Bigda J, Szymanski M. Effectiveness of Tranexamic Acid in Reducing Hidden Blood Loss During Laparoscopic Sleeve Gastrectomy: A Randomized Clinical Trial. J Clin Med. 2025 Apr 26;14(9):3010. doi: 10.3390/jcm14093010. PMID 40364042
- [Background] Lech P, Michalik M, Waczynski K, Osowiecka K, Dowgiallo-Gornowicz N. Effectiveness of prophylactic doses of tranexamic acid in reducing hemorrhagic events in sleeve gastrectomy. Langenbecks Arch Surg. 2022 Nov;407(7):2733-2737. doi: 10.1007/s00423-022-02630-5. Epub 2022 Aug 3. PMID 35920900
- [Background] Brito RM, Oliveira CMB, Moura ECR, Campelo GP, Lima RC, Fe CSM, Sousa TM, Oliveira EJSG, Dibai Filho AV, Leal PDC. Tranexamic acid effects in postoperative bleeding outcomes in laparoscopic sleeve gastrectomy: a controlled study. Acta Cir Bras. 2022 Oct 10;37(7):e370702. doi: 10.1590/acb370702. eCollection 2022. PMID 36228297